CLINICAL TRIAL: NCT06553950
Title: Mandibular Splint Versus Botox Injection in Lateral Pterygoid on Cervical Muscle Activity in Patients With Temporomandibular Disorders
Brief Title: Mandibular Splint vs Botox Injection in Lateral Pterygoid on Cervical Muscle Activity in Patients With Temporomandibular Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kerolos Ghobrial Goda Abd-El Malak, Resident of Physical Therapy , Faculty of Physical Therapy ,Cairo University, Cairo, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004426
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Mandibular Splint; Botox; Lateral Pterygoid; Cervical Muscle Activity; Temporomandibular Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Botox injection group (Experimental): Patients will be treated by Botox injection in lateral pterygoid muscle and medications like muscle relaxants, antidepressants, and nonsteroidal anti-inflammatory drugs.
  A Botox-A vial was diluted with normal saline to a concentration of 10 U per 0.1 mL for injection in a 1-ml insulin syringe. This will be injected into the ipsilateral lateral pterygoid muscle
  Interventions: Drug: Botox injection
- Mandibular stabilization splint group (Experimental): Patients will be treated by mandibular stabilization splint and medications like muscle relaxants, antidepressants and nonsteroidal anti-inflammatory drugs.
  Interventions: Drug: Mandibular stabilization splint
- Control group (Active Comparator): Patients will be treated by medications like muscle relaxants, antidepressants and nonsteroidal anti-inflammatory drugs.
  Interventions: Drug: Muscle relaxant

INTERVENTIONS:
Drug: Botox injection — Patients will be treated by Botox injection in lateral pterygoid muscle and medications like muscle relaxants, antidepressants and nonsteroidal anti-inflammatory drugs.
  A Botox-A vial was diluted with normal saline to a concentration of 10 U per 0.1 mL for injection in a 1-ml insulin syringe. This will be injected into the ipsilateral lateral pterygoid muscle.
  Arms: Botox injection group
Drug: Mandibular stabilization splint — Patients will be treated by mandibular stabilization splint and medications like muscle relaxants, antidepressants and nonsteroidal anti-inflammatory drugs.
  Arms: Mandibular stabilization splint group
Drug: Muscle relaxant — Patients will be treated by medications like muscle relaxants, antidepressants and nonsteroidal anti-inflammatory drugs.
  Arms: Control group

SUMMARY:
The study aims to compere mandibular splint versus botox injection in lateral pterygoid on cervical muscle activity in patients with temporomandibular disorders

DETAILED DESCRIPTION:
Temporomandibular disorders (TMD) are common chronic musculoskeletal pain conditions among orofacial pain, consisting of a group of conditions associated with pain and dysfunction of the temporomandibular joint (TMJ) and masticatory muscles. Temporomandibular joint displacement, also known as internal disc derangement, is an abnormal relationship between the articular disc, the mandibular condyle, and the mandibular fossa. The most frequent displacement of the disc is anterior to the mandibular condyle however, in rare cases it can be posteriorly.

Occlusal splint treatment is generally considered to be a basic treatment for Temporomandibular disorders. It could promote correction of the vertical dimension, maxillo-mandibular realignment, temporomandibular joint repositioning and cognitive awareness. Although various splints are currently available, the most used are stabilization splints and anterior repositioning splints.

Injection of BTX-A in LP muscle, considering the different methods, frequencies and injection dosages used in different studies, would decrease the clicks and other TMJ-related disorders such as pain, hyperactivity, and dysfunction. Based on the present review, most studies about the injection of botulinum toxin in LP muscle reported cases or were done as quasi-experimental studies.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18-40 years old.
* Both sexes.
* Duration of the disease is more than 3 months.
* Anterior mandibular disc displacement with reduction will be included.
* Unilateral anterior mandibular displacement with reduction grade 2&3 (Wilkes) will be included.
* Patients with cervical muscles spasm and trigger points (upper trapezius& sternocleidomastoid) will be included.
* Patients with sufficient cognitive abilities that enables them to understand and follow instructions.

Exclusion Criteria:

* Neurological or musculoskeletal diseases that affect cervical spine other than mandibular disc displacement (eg: cervical spondylosis, spondylolisthesis, and cervical disc injuries)
* Bilateral anterior mandibular disc displacement patients.
* Musculoskeletal disorders such as severe arthritis, cervical spine surgery or contractures of fixed deformity, leg length discrepancy.
* women during pregnancy and lactation.
* Patients with known hypersensitivity to any component of the drug (especially hypersensitivity to human albumin).
* Patients with infection or inflammation of the area where the toxin injections are planned, in patients with musculoskeletal conduction disorders, in primary muscular disorders (muscular dystrophy, neuromyopathy, congenital myopathies, myotonic disorders, mitochondrial myopathy and unspecified or other primary muscle disorders).
* Patients being treated with aminoglycoside antibiotics, ciclosporin, D-penicillamine, tubocurarine, pancuronium, gallamine, succinylcholine, chloroquine, or hydroxychloroquine.
* History of cervical spine surgery.
* History of trauma or fractures in cervical spine.
* Signs of cervical radiculopathy or myelopathy.
* Vascular syndrome such as vertebrobasilar insufficiency.
* Signs of serious pathology ( e.g., malignancy, inflammatory disorders, infection).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Muscle activity of upper trapizieus and sternocleidomastoid | After injection for 3 months.
  Muscle activity of upper trapizieus and sternocleidomastoid will be recorded before and after injection for 3 months by neurosoft Electromyography

SECONDARY OUTCOMES:
Amplitude of muscle activity | After injection for 3 months.
  Amplitude of muscle activity will be recorded before and after injection for 3 months by neurosoft Electromyography.
Root mean square of muscle activity | After injection for 3 months.
  Root mean square of muscle activity will be recorded before and after injection for 3 months by neurosoft Electromyography.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.